CLINICAL TRIAL: NCT02626520
Title: Phase 2 Evaluation of a Community-Based Multi-modality Management Algorithm for Clinically Non-metastatic Ductal Adenocarcinoma of the Exocrine Pancreas or Ampulla
Brief Title: Phase 2 Evaluation of Multi-modality Algorithm for Non-metastatic Adenocarcinoma of Pancreas or Ampulla
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study team felt toxicity of study regimen outweighed potential benefit.
Sponsor: Essentia Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PANC-1
Record Dates: First submitted 2015-12-03; First posted 2015-12-10 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-10

CONDITIONS: Ductal Adenocarcinoma of Pancreas; Adenocarcinoma of Ampulla
MeSH Terms: interventions — Gemcitabine; Taxes; Fluorouracil; Irinotecan; Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resectable, Low Risk (Experimental): Systemic chemotherapy followed by definitive surgery without pre-operative or post-operative radiotherapy.
  Interventions: Drug: Gemcitabine and nanoparticle albumin bound paclitaxel; Procedure: Definitive resection
- Locally Advanced (Experimental): Systemic chemotherapy followed by chemoradiation, followed by definitive surgery
  Interventions: Drug: Gemcitabine and nanoparticle albumin bound paclitaxel; Drug: 5-fluorouracil and irinotecan; Radiation: Preoperative chemoradiation; Procedure: Definitive resection

INTERVENTIONS:
Drug: Gemcitabine and nanoparticle albumin bound paclitaxel — Gemcitabine and nab-paclitaxel given every 14 days x 4 cycles
  Other Names: Gem/Abraxane, Gemcitabine/nab-paclitaxel
Drug: 5-fluorouracil and irinotecan — FOLFIRI.3 given every 14 days x 4 cycles
  Other Names: FOLFIRI.3, FOLFIRI-3
  Arms: Locally Advanced
Radiation: Preoperative chemoradiation — Pre-operative chemoradiation to 40 Gy in 20 fractions
  Arms: Locally Advanced
Procedure: Definitive resection — Definitive surgical resection of primary tumor
  Other Names: pancreaticoduodenectomy, Whipple procedure

SUMMARY:
Patients diagnosed with pancreatic cancer without clinically detectable metastatic disease will be treated with standardized systemic chemotherapy, followed by chemoradiation, and then surgical resection for those with resectable or borderline resectable disease. The primary endpoint is disease-free survival at 1 yr from initiation of treatment.

DETAILED DESCRIPTION:
Patients with ductal adenocarcinoma of the pancreas (or ampulla) that have received no prior therapy and have no clinically detectable metastatic disease will be enrolled. Management will be driven by resectability status as defined by the American College of Surgeons. All patients will be defined at entry as Resectable, Borderline Resectable or Locally Advanced (Unresectable).

All patients will be treated initially with gemcitabine and nanoparticle albumin bound paclitaxel (nab-paclitaxel) every 14 days for 4 cycles. Patients classified as Resectable, who have CA19-9 below 180 and CA-125 below 30 will then proceed to resection. All other patients will get 5-fluorouracil as 46 hr infusion given with leucovorin and irinotecan (FOLFIRI-3) every 14 days x 4 cycles.

All patients without progression will then receive chemoradiation consisting of external beam radiotherapy (40 Gy in 20 fractions given over 4 weeks). During radiation all patients will receive radiosensitizing radiotherapy as: 5-fluorouracil at 225 mg/m2 5 days per week, Mitomycin-C at 3 mg.m2 on d1, 8, 15 & 22; Cisplatin at 10 mg/m2 on d2, 9, 16, 23 and unfractionated heparin at 6,000 units/m2 daily in divided doses from day 1 to day 28.

After approximately 4 weeks to recover from chemoradiation, all patients with Resectable or Borderline Resectable disease will undergo definitive surgery.

Adjuvant therapy with FOLFIR-3 for an additional 6 cycles will be offered to all patients post-operatively.

Patients will then be actively followed every 3 to 6 months in keeping with National Comprehensive Cancer Network (NCCN) guidelines for 2 yrs, and then followed for recurrence, late toxicity and vital status every 6 months through 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of adenocarcinoma consistent with ductal carcinoma of pancreas or ampulla, with no evidence of metastatic disease by clinical exam or cross-sectional imaging.
* Fitness for chemotherapy in judgement of treating physician
* Bilirubin < 4 (any means of biliary drainage acceptable)

Exclusion Criteria:

* Medical or mental illness precluding provision of informed consent
* Pregnancy
* Active infection for which neutropenia would pose high risk of mortality

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kebbekus, MD, PhD, Principal Investigator — Essentia Health Cancer Center
Locations (1):
- Essentia Health Cancer Center, Duluth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make unidentified dataset available for electronic download.

REFERENCES:
- Available data/document: Study Protocol — https://docs.google.com/viewer?a=v&pid=sites&srcid=ZGVmYXVsdGRvbWFpbnxyZWFsd29ybGRvbmNvbG9neXxneDo2OGI0ZDgxMzdkZDIxYWJh

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Resectable, Low Risk | Locally Advanced
Started | 1 | 10
Completed | 0 | 0
Not Completed | 1 | 10
Not completed — Physician Decision | 1 | 1
Not completed — Adverse Event | 0 | 4
Not completed — Lack of Efficacy | 0 | 2
Not completed — Did not start protocol therapy | 0 | 2
Not completed — Study terminated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resectable, Low Risk | Locally Advanced | Total
Number analyzed (Participants) | 1 | 10 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 7 | 8
  >=65 years | 0 | 3 | 3
Age, Continuous [Median (Full Range); unit: years] | 64 [64 to 64] | 63 [57 to 80] | 63 [57 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 0 | 4 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 10 | 11

OUTCOME MEASURES:

1. Primary Outcome: Relapse Free Survival
Description: Percentage of patients alive and free of detectable disease 1 yr from start of treatment
Time Frame: 1 yr form onset of treatment
Population: Due to excessive toxicity of study regimen, the study was permanently closed prior to data analysis.
Arm/Group | Resectable, Low Risk | Locally Advanced
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: R-0 Rate
Description: Rate of patients having surgery who have negative surgical margins (i.e. R-0 resection)
Time Frame: Time of surgery
Population: Data not collected, study Terminated
Arm/Group | Resectable, Low Risk | Locally Advanced
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival
Description: Time to death from any cause measured from start of treatment
Time Frame: Up to 3 years from registration
Population: Data not collected, study terminated
Arm/Group | Resectable, Low Risk | Locally Advanced
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study enrollment through study termination, on average approximately 3 months
Arm/Group | Resectable, Low Risk | Locally Advanced
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/10
Serious Adverse Events (participants affected / at risk) | 0/1 | 3/10
Other Adverse Events (participants affected / at risk) | 0/1 | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resectable, Low Risk (N=1) | Locally Advanced (N=10)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resectable, Low Risk (N=1) | Locally Advanced (N=10)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No